CLINICAL TRIAL: NCT04891354
Title: A Single-Blind, Placebo-Controlled, First-in-Human Study to Assess the Safety and Tolerability of PDNO Administered as an Intravenous Infusion in Healthy Subjects
Brief Title: A First-in-Human Study to Assess the Safety and Tolerability of PDNO
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Attgeno AB (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-PDNO-001
Record Dates: First submitted 2021-05-06; First posted 2021-05-18 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Pulmonary Hypertension
Keywords: Acute Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — 1-(nitrosooxy)propan-2-ol and 2-(nitrosooxy)propan-1-ol drug combination; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: In Part I, each subject will receive a 30 minute i.v. infusion of placebo followed by a 1-hour i.v. infusion of PDNO in parallel with a carrier sodium bicarbonate buffer, the infusion of which will start 5 minutes prior to start of placebo infusion and continue until 15 minutes after end of PDNO infusion. Between the end of placebo infusion and prior to the start of PDNO infusion, there will be a 20-minute stabilisation period with infusion of sodium bicarbonate buffer only.
  In Part II, each subject will receive a 30 minute i.v. infusion of placebo followed by 2 x 30 minute infusions of PDNO at 2 ascending dose levels and one 3-hour infusion of PDNO at a third dose level.
Who Masked: Participant
Masking Description: During the administration, the infusion set is masked for the subject.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part I: single ascending dose (SAD) (Experimental): In Part I, each subject will receive a 30 minute i.v. infusion of placebo followed by a 1-hour i.v. infusion of PDNO in parallel with a carrier sodium bicarbonate buffer, the infusion of which will start 5 minutes prior to start of placebo infusion and continue until 15 minutes after end of PDNO infusion. Between the end of placebo infusion and prior to the start of PDNO infusion, there will be a 20-minute stabilisation period with infusion of sodium bicarbonate buffer only.
  Interventions: Drug: PDNO; Drug: Sodium chloride (placebo)
- Part II: ascending doses of PDNO (Experimental): In Part II, each subject will receive a 30 minute i.v. infusion of placebo followed by 2 x 30 minute infusions of PDNO at 2 ascending dose levels and one 3-hour infusion of PDNO at a third dose level.
  Interventions: Drug: PDNO; Drug: Sodium chloride (placebo)

INTERVENTIONS:
Drug: PDNO — PDNO consists of propylene glycol (1,2-propanediol, PD) chemically combined with NO (to be donated). The drug substance is formulated as an inherent mixture of 4 structure analogues. The mixture consists of an equilibrium of the 2 regioisomers 1-(nitrosooxy) propan-2-ol and 2-(nitrosooxy) propan-1-ol. In addition, each regioisomer is a racemic mixture.
  Other Names: Nitrosooxypropanol
Drug: Sodium chloride (placebo) — Placebo (NaCl, commercially available dilution solution for parenteral use, 9 mg/mL)
  Other Names: NaCl

SUMMARY:
This is a first-in-human, single-blind, placebo-controlled, single-centre study designed to assess the safety and tolerability of PDNO in healthy male and female subjects. In addition, the exposure of 1,2 propanediol (PD) will be evaluated.

There are 2 parts to the study:

Part I: single ascending dose (SAD), 7 cohorts, 30 minutes intravenous (i.v.) infusion of placebo followed by 1-hour i.v. infusion of PDNO to assess safety, tolerability and PD exposure in healthy male and female subjects.

Part II: ascending doses of PDNO in 2 cohorts, 30 minutes i.v. infusion of placebo followed by 3 ascending doses of PDNO in cohort 1 and 3 ascending doses of PDNO in cohort 2. The first 2 doses in each cohort will be i.v. infused for 30 minutes whereas the last will be i.v. infused for 3 hours to assess safety, tolerability and PD exposure in healthy male and female subjects.

If indicated by emerging data and recommended by the internal safety review committee (iSRC), 2 additional dose groups/cohorts (4+4 subjects) may be added to Part I and 1 dose group/cohort (4 subjects) may be added to Part II.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give written informed consent for participation in the study
* Healthy male and female subjects aged 18 to 45 years inclusive at screening
* Body Mass Index (BMI) ≥ 18.5 and ≤ 30.0 kg/m^2 at screening
* Clinically normal medical history, physical findings, ECG and laboratory values
* Male subjects and women of non-childbearing potential may be included in the study. Male subjects must be willing to use condom or be vasectomised or practice sexual abstinence to prevent pregnancy and drug exposure of a female partner and refrain from donating sperm from the date of dosing until 3 months after dosing with the IMP. Their female partner of child-bearing potential must use contraceptive methods.
* Women of non-childbearing potential are defined as pre-menopausal females who are sterilised or postmenopausal

Exclusion Criteria:

* History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, might interfere with the drug absorption, distribution, metabolism or excretion of the drug or influence the results or the subject's ability to participate in the study
* Any clinically significant illness, medical/surgical procedure or trauma within 4 weeks of the first administration of IMP
* Malignancy within the past 5 years
* Any planned major surgery within the duration of the study
* Any positive result on screening for serum hepatitis B surface antigen, hepatitis C antibody and Human Immunodeficiency Virus (HIV)
* Women who are pregnant or who are breast feeding
* Known patent foramen ovale or other cardiac phenomenon putting the subject at risk in the study
* Presence of history of Raynaud Syndrome
* After 10 minutes supine rest at the time of screening, any vital sign values outside the following ranges: Systolic blood pressure <90 or >140 mmHg, or Diastolic blood pressure <50 or >90 mmHg, or Pulse <40 or >90 bpm
* Prolonged QTcF (>450 ms), cardiac arrhythmias or any clinically significant abnormalities in the resting ECG at the time of screening, as judged by the Investigator
* Known history of migraine or frequent headache of other genesis (in average >1 episode of grade 2 (CTCAE v5.0, headache per week)
* History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the Investigator, or history of hypersensitivity to drugs with a similar chemical structure or class to PDNO
* History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity to the local anaesthesia planned to be used in the study
* Known hypersensitivity to propanediol
* Veins unsuitable for CVC and arterial cannula insertion
* Failure to perform the FeNO measurement at screening
* FeNO level ≥ 30 ppb
* Within 1 month prior to Screening received continuous treatment with non-steroidal anti-inflammatory drugs (NSAIDs), novel oral anticoagulants (NOACs), warfarin, clopidogrel, or acetylsalicylic acid
* Regular use of any prescribed or non-prescribed medication including antacids, analgesics, herbal remedies, vitamins and minerals within 2 weeks prior to the (first) administration of IMP
* Planned treatment or treatment with another investigational drug within 3 months prior to Day -1
* Current smokers or users of nicotine products
* Positive screen for drugs of abuse or alcohol
* Presence or history of alcohol abuse or excessive intake of alcohol
* Presence or history of drug abuse, as judged by the Investigator
* History of, or current use of, anabolic steroids
* Excessive caffeine consumption defined by a daily intake of >5 cups of caffeine containing beverages
* Intake of xanthine and/or taurine containing energy drinks at the day of screening.
* Plasma donation within one month of screening or blood donation
* Investigator considers the subject unlikely to comply with study procedures, restrictions and requirements
* Previous confirmed COVID-19 that required hospitalisation
* Signs or symptoms probably consistent with COVID-19 disease within the last 7 days prior to Visit 2 or close contact with confirmed COVID-19 patient within the last 7 days prior to Visit 2, as judged by the Investigator
* Positive result for ongoing SARS-CoV-2 presented at Visit 2

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2021-02-02 (Actual); Primary Completion 2022-05-25 (Actual); Study Completion 2022-05-25 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of PDNO following i.v. infusion to healthy volunteers, as measured by incidence of treatment-emergent AEs, SAEs, AESI, changes in vital signs, ECG abnormalities, and laboratory abnormalities. | Through study completion (i.e., Day 8)
  * Treatment-emergent adverse events (AEs)
  * Treatment-emergent serious AEs (SAEs)
  * Treatment-emergent AEs of special interest (AESI)
  * Treatment-emergent changes in vital signs (blood pressure, pulse, oxygen saturation, respiratory frequency, body temperature)
  * Treatment-emergent electrocardiogram (ECG) abnormalities
  * Treatment-emergent laboratory abnormalities

SECONDARY OUTCOMES:
Exposure parameters for 1,2-propanediol (PD): area under the curve from time 0 to time t (AUC0-t) | During 24 hours from start of dosing
Exposure parameters for 1,2-propanediol (PD): area under the curve from time 0 to infinity (AUC0-inf) | During 24 hours from start of dosing
Exposure parameters for 1,2-propanediol (PD): maximum plasma concentration (Cmax) | During 24 hours from start of dosing
Exposure parameters for 1,2-propanediol (PD): terminal elimination half-life (T1/2) | During 24 hours from start of dosing

OTHER OUTCOMES:
Change in FeNO levels before and after i.v. infusion of PDNO | During Day 1
  FeNO levels (Part 1 only) as measured using a NIOX VERO airway inflammation monitor.
Collection of plasma for future analysis of biomarkers such as nitrite and nitrate in plasma (µM) | During Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Folke Sjöberg, MD, Principal Investigator — CTC Clinical Trial Consultants AB
Locations (1):
- CTC Clinical Trial Consultants AB, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No